CLINICAL TRIAL: NCT05965973
Title: Short-term Impact of a Low Carbohydrate/high Unsaturated Fat Diet on Hepatic Transcriptomics and Lipidomics in Individuals with Pre-diabetes - a Pilot Study
Brief Title: Diet Impact on Hepatic Transcriptomics and Lipidomics in Pre-diabetes
Acronym: DGENE-NAFLD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Couture, MD, PhD, FRCP (C), Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: INAF 2023-6814
Record Dates: First submitted 2023-06-12; First posted 2023-07-28 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Diet, Fat-Restricted; Diet, High-Fat

STUDY DESIGN:
Who Masked: Participant
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low fat diet (Experimental): During 3 days, subjects eat a diet low in fat (percent of total caloric intake: 15.0% from proteins; 65.0% from carbohydrates; 20.0% from fat: 4.0% from saturated fat; 10.0% from monounsaturated fat; 6.0% from polyunsaturated fat
  Interventions: Other: Low fat diet; Other: High fat diet
- High fat diet (Experimental): During 3 days, subjects eat a diet high in fat (percent of total caloric intake: 15.0% from proteins; 45.0% from carbohydrates; 40.0% from fat: 8.0% from saturated fat; 22.0% from monounsaturated fat; 10.0% from polyunsaturated fat
  Interventions: Other: Low fat diet; Other: High fat diet

INTERVENTIONS:
Other: Low fat diet — During 3 days, subjects eat a diet low in fat (percent of total caloric intake: 15.0% from proteins; 65.0% from carbohydrates; 20.0% from fat: 4.0% from saturated fat; 10.0% from monounsaturated fat; 6.0% from polyunsaturated fat
Other: High fat diet — During 3 days, subjects eat a diet high in fat (percent of total caloric intake: 15.0% from proteins; 45.0% from carbohydrates; 40.0% from fat: 8.0% from saturated fat; 22.0% from monounsaturated fat; 10.0% from polyunsaturated fat

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is one of the most common liver diseases, affecting 25% to 30% of the global population and nearly one third of the population in North America. NAFLD is defined as an excessive accumulation of lipids within hepatocytes in the absence of significant alcohol consumption or other causes of chronic liver disease. These patients usually present with hepatic steatosis observed on imaging studies and elevated liver enzymes with clinical features of insulin resistance (IR), including pre-diabetes, type 2 diabetes mellitus (T2DM), arterial hypertension, dyslipidemia, and visceral obesity. The minimum criterion for a histologic diagnosis of NAFLD is >5 percent steatotic hepatocytes in a liver tissue section. The exact mechanism for the development of NAFLD is unclear, although the current evidence indicates that it is likely a complex interplay among neurohormones, intestinal dysbiosis, nutrition, and genetics. IR plays a crucial role in NAFLD pathophysiology mainly by increasing adipocyte lipolysis, resulting in the circulation of more free fatty acids available for hepatic uptake and increasing hepatic de novo lipogenesis. There is yet no approved pharmacologic option for the treatment of NAFLD. Current international guidelines on NAFLD emphasize the importance of lifestyle modifications for all patients with NAFLD and recommend 7-10% of weight loss and a "healthy diet", without suggesting any particular diet. Recent data provide some support for the beneficial role of low carbohydrate (CHO)/high unsaturated fatty acid (both monounsaturated (MUFAs) and polyunsaturated (PUFAs)) dietary patterns for decreasing hepatic steatosis. This proposal addresses this important research gap by leading to advances regarding the impact of a short-term low CHO/high PUFAs/MUFAs dietary intervention on improving hepatic gene expression profiles and lipid composition in individuals with pre-diabetes. The proposed study is unique because all meals and foods will be provided to participants under carefully controlled isocaloric conditions to maintain a constant bodyweight with optimal energy and macronutrient intake control. The primary objective of the proposed research is to investigate how replacement of dietary CHOs by unsaturated fatty acids (both PUFAs and MUFAs) affects liver fat composition and liver transcriptomics in subjects with pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 60 years of age.
* Non-smoker
* Waist circumference > 102 cm for men and > 88 cm for women.
* Plasma triglyceride levels > 1,7 mmol/L at the screening visit.
* Fasting plasma glucose levels > 6,1 mmol/L at the screening visit.
* Fasting plasma insulin levels above the upper limit of normal at the screening visit.
* Subjects must be willing to give written informed consent and able to adhere to the diet schedule and visit schedule.
* Patients should be otherwise healthy, without abnormal renal function or coagulation.

Exclusion Criteria:

* Patients with extreme dyslipidemias, such as familial hypercholesterolemia will be excluded.
* Subjects will be excluded if they have cardiovascular disease (CHD, cerebrovascular disease or peripheral arterial disease) or if they are taking other medications known to affect lipoprotein metabolism (eg. steroids, beta blockers, thiazide diuretics, other lipid lowering agents, significant alcohol intake etc.).
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Individuals with a history of mental instability, drug or alcohol abuse within the past 2 years or individuals who have been treated or are being treated for severe psychiatric illness that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Disorders of the hematologic, digestive, or central nervous systems, including cerebrovascular disease and degenerative disease, that would limit study evaluation or participation.
* Known impairment of renal function (creatinine >2.0 mg/dL), dysproteinemia, nephrotic syndrome, or other renal disease.
* Subjects with coagulopathy (prothrombin time [PT] or partial thromboplastin time [PTT] at Visit 1 higher than 1.5 times control).
* Patients who are known to have tested positive for human immunodeficiency virus (HIV).
* Patients who have used any investigational drug within 30 days of the first clinic visit.
* Diabetic patients are excluded from the study. Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins. Clinically euthyroid subjects on replacement doses of thyroid hormone are eligible for enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the expression of key genes in lipid metabolism including LDL-receptor, acetyl-CoA acetyltransferase 2, apolipoprotein B, proproprotein convertase subtilisin/kexin type 9, microsomal triglyceride transfer protein | At Day 3 and day 20 (at the end of the two 3-day diets)
Change in the expression of key genes in liver inflammation including C-reactive protein, Interleukin-6, Interleukin-15, cell adhesion molecules, E-selectin | At Day 3 and day 20 (at the end of the two 3-day diets)
Change in the expression of key genes in hepatic fibrogenesis including transforming growth factor beta 1, a-smooth muscle actin, type-1 collagen, connective tissue growth factor | At Day 3 and day 20 (at the end of the two 3-day diets)

SECONDARY OUTCOMES:
Change in liver's key lipid pathways (lipidomics) including lysophosphatidylcholine, phosphatidylcholine, diglyceride. | At Day 3 and day 20 (at the end of the two 3-day diets)
Identify bacteria strains involved in the control of blood glucose such as C elegans. | At Day 3 and day 20 (at the end of the two 3-day diets)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada